CLINICAL TRIAL: NCT06414616
Title: Are We Overly Concerned About Rebound Fractures? Real-World Evidence of Adherence to Denosumab Therapy and Fracture Risk Associated With Drug Withdrawal: A Cross-sectional Study
Brief Title: Real-World Evidence of Adherence to Denosumab Therapy and Fracture Risk Associated With Drug Withdrawal: A Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Hande Ozdemir, Assoc. Prof., Trakya University
Other Study IDs: 2022/343
Record Dates: First submitted 2022-12-06; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Osteoporosis
Keywords: Denosumab; Fragility fracture; Rebound fracture; Discontinuation; Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the light of current literature data, it is not recommended to discontinue Denosumab therapy without initiating another antiresorptive therapy. It is known that there is a rebound increase in bone resorption markers and a rapid decrease in bone mineral density (BMD) when patients using Denosumab remain untreated for 1 year. The coronavirus disease (Covid-19) pandemic has caused an unprecedented disruption in the management of osteoporosis, as in many chronic diseases. This study aims to determine whether the risk of rebound-associated osteoporotic fracture development is increased in patients who discontinued Denosumab therapy due to any reason but especially due to hesitancy to come to hospitals or lack of access to treatment institutions during the pandemic period as well as to evaluate the factors affecting treatment compliance.

DETAILED DESCRIPTION:
With increased life expectancy and decreased physical activity osteoporosis related fractures are increasing day by day which place a huge health economic burden on societies. Since fragility fractures and related disabilities bring about considerable morbidity and even mortality, the main goal in osteoporosis treatment is to prevent fractures.

The facts that bisphosphonates can plateau after 3-4 years in the treatment response and Teriparatide cannot be used for more than 2 years, bring the use of Denosumab to the fore in patients with high fracture risk who need long term treatment. Denosumab is also preferred in patients with renal dysfunction since it is excreted by the reticuloendothelial system and not the kidney. However, there is a dilemma that publications in the literature mostly show that the risk of fracture development returns to a no-treatment status shortly after Denosumab withdrawal.

Therefore, in this study it is aimed to examine whether there is statistically significant difference in terms of the risk of osteoporotic fracture development and other secondary outcome measures between the patient group who discontinued injections for more than 2 months and the patient group who regularly received their injections.

In this study, patients who had commenced Denosumab in Trakya University Osteoporosis Polyclinic between 2015-2021 and had received at least 2 doses will be included. Demographic and clinical data will be retrospectively examined by the Physical Medicine and Rehabilitation physician at last date of follow-up through electronic medical records and patient files. Radiological images of the patients will also be examined whether there is radiological fracture before, under or after the treatment. The number of fractures and their localizations, if any, will be recorded. The number of Denosumab doses administered will be determined by review of the hospital's electronic prescription records. Adherence will be defined as being punctual (with an allowable delay of up to 8 weeks) with the 6 month scheduled doses. In addition, pre-treatment values of BMD as evaluated on dual energy x-ray absorptiometry (DXA), and Fracture Risk Assessment Tool (FRAX) scores will be recorded.

In the light of the data obtained, the parameters affecting compliance and the effect of treatment compliance on the risk of osteoporotic fracture development will be presented to the literature.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients who had received at least two consecutive doses of Denosumab ,with a gap of fewer than 8 months, with the diagnosis of osteoporosis.
* 2. Patients who had at least one radiological image before the initiation of Denosumab therapy in which the lumbar and thoracic spine could be visualised
* 3. Patients whose BMD and T-score values had been evaluated via DXA scan and FRAX scores had been calculated before the initiation of Denosumab therapy.

Exclusion Criteria:

* 1. Patients missing any of the above mentioned data
* 2. Patients who develop fractures due to cancer, trauma or Paget's disease.
* 3. Patients receiving monthly Denosumab to prevent bone metastasis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients initiated on Denosumab therapy at Trakya University Pyhsical Medicine and Rehabilitation Osteoporosis Unit between 2015-2021 and had received at least 2 doses of injection.
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Number of new fragility fractures | Through study completion, an average of 2 years
  The number of new fragility fractures among Denosumab adherent and non-adherent patient groups as assessed by radiological images

SECONDARY OUTCOMES:
Denosumab adherence rate and factors that may play a role in Denosumab adherence/non-adherence | Through study completion, an average of 2 years
  The rate of Denosumab adherence and factors that may play a role in Denosumab adherence/non-adherence as assessed by restrospective examination of patient files which are age, sex, age of menopause, parity, marital status, occupation, height (cm), weight (kg), and body mass index (BMI) (kg/m2), family history of fragility fracture, presence of baseline fragility fractures before initiation of Denosumab treatment, comorbidities, use of steroids, smoking status, presence of secondary osteoporosis, tea/coffee/alcohol consumption status, consumption of dairy products, presence of any therapy before Denosumab, treatment agent before Denosumab, number of received Denosumab injections, duration of Denosumab withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Hande Özdemir, MD, Principal Investigator — Trakya University
Locations (1):
- Trakya University Medical Faculty, Edirne, Turkey (Türkiye)

REFERENCES:
- [Background] Lyu H, Jundi B, Xu C, Tedeschi SK, Yoshida K, Zhao S, Nigwekar SU, Leder BZ, Solomon DH. Comparison of Denosumab and Bisphosphonates in Patients With Osteoporosis: A Meta-Analysis of Randomized Controlled Trials. J Clin Endocrinol Metab. 2019 May 1;104(5):1753-1765. doi: 10.1210/jc.2018-02236. PMID 30535289
- [Background] Brown JP, Roux C, Torring O, Ho PR, Beck Jensen JE, Gilchrist N, Recknor C, Austin M, Wang A, Grauer A, Wagman RB. Discontinuation of denosumab and associated fracture incidence: analysis from the Fracture Reduction Evaluation of Denosumab in Osteoporosis Every 6 Months (FREEDOM) trial. J Bone Miner Res. 2013 Apr;28(4):746-52. doi: 10.1002/jbmr.1808. PMID 23109251
- [Background] Black DM, Schwartz AV, Ensrud KE, Cauley JA, Levis S, Quandt SA, Satterfield S, Wallace RB, Bauer DC, Palermo L, Wehren LE, Lombardi A, Santora AC, Cummings SR; FLEX Research Group. Effects of continuing or stopping alendronate after 5 years of treatment: the Fracture Intervention Trial Long-term Extension (FLEX): a randomized trial. JAMA. 2006 Dec 27;296(24):2927-38. doi: 10.1001/jama.296.24.2927. PMID 17190893
- [Background] Sosa-Henriquez M, Torregrosa O, Deniz A, Saavedra P, Ortego N, Turrion A, Perez Castrillon JL, Diaz-Curiel M, Gomez-Alonso C, Martinez G, Antonio Blazquez J, Olmos-Martinez JM, Etxebarria I, Caeiro JR, Mora-Pena D. Multiple vertebral fractures after suspension of denosumab. A series of 56 cases. Int J Clin Pract. 2021 Oct;75(10):e14550. doi: 10.1111/ijcp.14550. Epub 2021 Jun 30. PMID 34145944
- [Background] Anastasilakis AD, Evangelatos G, Makras P, Iliopoulos A. Rebound-associated vertebral fractures may occur in sequential time points following denosumab discontinuation: need for prompt treatment re-initiation. Bone Rep. 2020 Apr 22;12:100267. doi: 10.1016/j.bonr.2020.100267. eCollection 2020 Jun. PMID 32373677
- [Background] Aubry-Rozier B, Gonzalez-Rodriguez E, Stoll D, Lamy O. Severe spontaneous vertebral fractures after denosumab discontinuation: three case reports. Osteoporos Int. 2016 May;27(5):1923-5. doi: 10.1007/s00198-015-3380-y. Epub 2015 Oct 28. PMID 26510845
- [Background] Niimi R, Kono T, Nishihara A, Hasegawa M, Kono T, Sudo A. Second rebound-associated vertebral fractures after denosumab discontinuation. Arch Osteoporos. 2020 Jan 2;15(1):7. doi: 10.1007/s11657-019-0676-0. PMID 31898803
- [Background] Fu SH, Wang CY, Hung CC, Lee CC, Yang RS, Huang CC, Farn CJ, Lin WH, Chen HM, Hsiao FY, Lin JW, Li CY. Increased fracture risk after discontinuation of anti-osteoporosis medications among hip fracture patients: A population-based cohort study. J Intern Med. 2021 Dec;290(6):1194-1205. doi: 10.1111/joim.13354. Epub 2021 Aug 2. PMID 34237171
- [Background] Cramer JA, Amonkar MM, Hebborn A, Altman R. Compliance and persistence with bisphosphonate dosing regimens among women with postmenopausal osteoporosis. Curr Med Res Opin. 2005 Sep;21(9):1453-60. doi: 10.1185/030079905X61875. PMID 16197664
- [Background] Chandran M, Hao Y, Kwee AK, Cheen MHH, Chin YA, Ng VYT. Adherence to dosing schedule of denosumab therapy for osteoporosis during COVID-19 lockdown: an electronic medical record and pharmacy claims database study from Asia. Osteoporos Int. 2022 Jan;33(1):251-261. doi: 10.1007/s00198-021-06085-0. Epub 2021 Aug 21. PMID 34417842
- [Background] Siris ES, Harris ST, Rosen CJ, Barr CE, Arvesen JN, Abbott TA, Silverman S. Adherence to bisphosphonate therapy and fracture rates in osteoporotic women: relationship to vertebral and nonvertebral fractures from 2 US claims databases. Mayo Clin Proc. 2006 Aug;81(8):1013-22. doi: 10.4065/81.8.1013. PMID 16901023
- [Background] Black DM, Delmas PD, Eastell R, Reid IR, Boonen S, Cauley JA, Cosman F, Lakatos P, Leung PC, Man Z, Mautalen C, Mesenbrink P, Hu H, Caminis J, Tong K, Rosario-Jansen T, Krasnow J, Hue TF, Sellmeyer D, Eriksen EF, Cummings SR; HORIZON Pivotal Fracture Trial. Once-yearly zoledronic acid for treatment of postmenopausal osteoporosis. N Engl J Med. 2007 May 3;356(18):1809-22. doi: 10.1056/NEJMoa067312. PMID 17476007